CLINICAL TRIAL: NCT06937684
Title: Oral Fluid Timing and Volume in Children Aged 1-8 Following Ambulatory Surgery: A Prospective Randomized Controlled Trial
Brief Title: Early Oral Fluid Intake in Children After Day Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E2-24-6970
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Anesthesia; Postoperative Nausea and Vomiting (PONV); Ambulatory Surgical Procedures
Keywords: Perioperative fasting; Ambulatory surgery; Pediatric postoperative care; Clear fluid intake; Postoperative nausea and vomiting (PONV); Pediatric anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized controlled trial. Participants will be randomly assigned to one of two groups to receive a maximum of 10 ml/kg of clear fluids either 1 hour (early group) or 2 hours (traditional group) after general anesthesia. Each participant will be assigned to only one group and will receive the intervention once.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor (the nurse responsible for evaluating postoperative vomiting) is blinded to the group assignments. No other study personnel, caregivers, or participants are masked in this trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Oral Intake Group (Group E) (Experimental): Patients in this group will receive a maximum of 10 ml/kg of clear fluids (e.g., water or clear fruit juice) starting at 1 hour after the completion of general anesthesia.
  Interventions: Behavioral: Early Oral Fluid Intake
- Traditional Oral Intake Group (Group T) (Active Comparator): Patients in this group will receive a maximum of 10 ml/kg of clear fluids (e.g., water or clear fruit juice) starting at 2 hours after the completion of general anesthesia.
  Interventions: Behavioral: Traditional Oral Fluid Intake

INTERVENTIONS:
Behavioral: Early Oral Fluid Intake — Participants receive clear fluids up to 10 ml/kg at 1 hour after anesthesia.
  Arms: Early Oral Intake Group (Group E)
Behavioral: Traditional Oral Fluid Intake — Participants receive clear fluids up to 10 ml/kg at 2 hours after anesthesia.
  Arms: Traditional Oral Intake Group (Group T)

SUMMARY:
This study investigates the safety and tolerability of early oral clear fluid intake in children aged 1-8 years undergoing elective outpatient non-gastrointestinal surgeries. Patients will be randomized to receive clear fluids either at 1 hour or 2 hours after general anesthesia. The goal is to determine whether earlier fluid intake increases the risk of postoperative vomiting (POV), or whether it can be safely tolerated in pediatric patients."

DETAILED DESCRIPTION:
This prospective, randomized controlled clinical trial aims to evaluate the safety and tolerability of early oral clear fluid intake in children aged 1 to 8 years undergoing elective, outpatient, non-gastrointestinal surgery under general anesthesia. Recent guidelines recommend reducing preoperative and postoperative fasting durations in children to enhance recovery and well-being. Early postoperative hydration has been associated with reduced opioid requirements, faster return to normal diet and ambulation, and shorter hospital stay, without increasing the risk of postoperative nausea and vomiting (PONV).

In this study, participants will be randomly assigned to one of two groups. Group E (early group) will receive up to 10 ml/kg of clear fluids (e.g., water, clear juice) one hour after the end of anesthesia, while Group T (traditional group) will receive the same amount two hours after anesthesia. Patients will be evaluated for readiness to drink based on recovery of consciousness, protective airway reflexes, and absence of nausea or vomiting. Fluid will be administered slowly and under strict supervision by experienced staff, with emergency equipment readily available.

The incidence of vomiting will be assessed using a modified 4-point scale. Additional outcome measures include tolerability of oral fluids, time to readiness for discharge, and incidence of delayed postoperative vomiting on postoperative days 1 and 3, assessed via phone interviews with caregivers. This study seeks to provide evidence-based guidance on the optimal timing and volume of clear fluid intake in pediatric patients following ambulatory minor surgical procedures, contributing to more flexible and patient-centered perioperative fasting protocols.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 and 8 years
* ASA Physical Status I or II
* Undergoing elective, outpatient, non-gastrointestinal surgery under general anesthesia
* Expected to be discharged on the same day
* Parent/guardian provides informed consent

Exclusion Criteria:

* Emergency surgeries
* History of gastrointestinal disorders
* History of aspiration or recurrent vomiting
* Children with neurodevelopmental delay
* Intraoperative complications requiring ICU admission
* Refusal of oral intake postoperatively

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability of Early Oral Clear Fluid Intake in Children | From end of anesthesia to discharge (approximately 3-4 hours postoperative)
  The number of pediatric participants who are able to tolerate clear oral fluids (up to 10 ml/kg) administered 1 hour after general anesthesia without experiencing vomiting, desaturation (SpO₂ < 94%), or other adverse events. Tolerability is defined as successful ingestion of the planned fluid volume without signs of intolerance such as nausea, vomiting, or clinical deterioration.

SECONDARY OUTCOMES:
Total Volume of Oral Fluids Tolerated | Within 1 and 2 hours post-anesthesia
  Amount of oral clear fluid (in ml/kg) successfully consumed by participants during the initial postoperative oral hydration attempt.
Incidence of Postoperative Vomiting | From end of anesthesia to discharge (within approximately 4 hours)
  Number of participants who experience vomiting after receiving oral clear fluids, as assessed using a 4-point modified vomiting scale from anesthesia end until discharge.
Incidence of Postoperative Vomiting on Day 1 and Day 3 | Postoperative day 1 and day 3
  Number of participants with parent-reported postoperative nausea assessed via structured telephone interviews conducted on postoperative day 1 and day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sever, Assoc Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No